CLINICAL TRIAL: NCT06218420
Title: Evaluation of Stereotactic Body Radiotherapy as a Bridge Therapy for Hepatocellular Carcinoma Patients Enlisted for Liver Transplantation
Acronym: TRANSRAD-01
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: APHP210358
Record Dates: First submitted 2023-12-04; First posted 2024-01-23 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-05

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatocellular carcinoma; liver transplantation; bridging treatment; stereotactic body radiation therapy
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with hepatocellular carcinoma enlisted for a liver transplant and eligible for SBRT (Other): All patients enrolled in the trial and responding to inclusion/exclusion criteria will receive SBRT (a high-precision technique allowing to deliver a precise high dose irradiation on moving intrahepatic lesions).
  Interventions: Radiation: Stereotactic Body Radiotherapy (SBRT)

INTERVENTIONS:
Radiation: Stereotactic Body Radiotherapy (SBRT) — Stereotactic Body Radiotherapy (SBRT) is a non-invasive alternative and potentially efficient treatment of single or bilocular HCC. However, SBRT has not been validated as bridging therapy before LT in a prospective study yet.

SUMMARY:
The aim of this trial is to carry out the first prospective multicentric study which evaluates the efficacy and the safety of SBRT in HCC patients enlisted for LT and not suitable for other bridging interventional treatments (RF or TACE).

The incidence of hepatocellular carcinoma (HCC) is increasing worldwide and is currently the first indication for Liver transplantation (LT). HCC patients access to LT is not only determined by the underlying liver function but also by the alpha-fetoprotein (aFP) score which allows to better identify patients with high risk of recurrence. LT is the best curative treatment as it can cure both the tumor and the underlying liver disease. However, the access to LT is limited due to organ shortage and preserved liver function for the majority of the patients with HCC. Bridging therapies, such as ablation by radiofrequency (RF) or microwaves, or trans-arterial chemoembolization (TACE), are carried out routinely to prevent the risk of tumor progression and drop-out during the waiting time (the drop-out rate being 20%). Nevertheless, only 50 to 70% of patients in France will have access to these treatments due to specific contraindications.

Stereotactic body radiotherapy (SBRT) has emerged as a non-invasive alternative and potentially efficient treatment of single or bilocular HCC. SBRT is a high-precision technique allowing to deliver a precise high dose irradiation on moving intrahepatic lesions. RTS is feasible only when the hepatic reserve is sufficient to avoid radic hepatitis.

Advantages of SBRT, as compared to TACE or RF, are 1) to preserve the hepatic artery, which can be altered by TACE 2) to allow access to complex tumors locations or superficial lesions not feasible by RF 3) to avoid any tumor spread related to punctures 4) to avoid general anesthesia.

However, SBRT has not been validated as bridging therapy before LT in a prospective study. Thus, this study is the first prospective multicentric study to evaluate this treatment modality in HCC patients enlisted for LT not suitable to RF or TACE.

DETAILED DESCRIPTION:
Hypothesis for the study:

The hypothesis is that SBRT in HCC patients enlisted for LT and not suitable to liver resection, RF, or TACE, is a safe and effective option to bring those patients to LT while limiting HCC progression during waiting time.

This study is the first prospective multicentric study to evaluate this treatment modality in this population.

Overview of the multimodal management of hepatocellular carcinoma Liver cancer is the fourth cause of cancer-related death (GLOBOCAN), with an increasing incidence over the last decades.

The best curative treatment for HCC remains liver transplantation (LT) as it can cure both the tumor and the underlying liver disease. 5-year survival rates reach 60-70% in patients with HCC after LT. However, the number of patients waiting for LT is by far exceeding the number of available donors: in 2017, there were 2.4 candidates for one graft (ABM, Rapport annuel). The global organ shortage and the risk of HCC recurrence after LT have therefore been taken into account in the therapeutic algorithm.

In France, patient's access to LT is determined by their liver function, assessed by the Model for End-stage Liver Disease (MELD) Score, which determines a national ranking on waiting list for LT depending on the severity of the liver impairment. The waiting list is managed by the National Biomédecine Agency (Agence de la Biomédecine). For HCC patients, the access to LT is not only determined by the underlying liver function but also by the alpha-fetoprotein (aFP) score, which allows to better identify patients with high risk of recurrence. An aFP Score ≤2 allows patient's access to LT by adding "HCC points" to the patient's national ranking calculation. HCC is currently the first indication for LT (32% of LT candidates in France).

Despite efforts are made to prioritize HCC patients on waiting list without disadvantaging other patients without HCC, the average waiting time for a LT remains 6 months and can go up to 12 months. Therefore, those patients face a significant risk of tumor progression during the waiting period, leading to tragic "drop-outs" from the waiting list, around 20-30% of patients with HCC. In this context, the transplant community has developed alternatives to prevent disease progression during the waiting period, referred to as "bridging therapies". It is recommended that patients who are expected to wait for more than 6 months for LT should be treated with bridging therapy.

The role of bridging therapies during waiting period for liver transplantation It has been demonstrated that reducing the amount of viable tumor in the liver improves the survival post-LT. The choice for one bridging therapy over others is made in expert multidisciplinary meetings depending on patient's characteristics, underlying liver function and HCC features and the range of bridging treatments proposed vary from potentially curative to palliative options (not curative). Up to date, no guidelines are available to decide which patients should receive bridging therapy. The American Association for the Study of Liver Diseases (AASLD) recommended subjecting every patient who is expected to wait for more than 6 months for LT to bridging therapies. In France, the proportion of patients receiving bridging therapies represents about 50 to 70% of patients enlisted for HCC.

The most frequent bridging therapies include Trans arterial Chemo embolization (TACE) and ablation (RF).

Focus on SBRT, an emerging therapy for HCC SBRT has emerged as a non-invasive alternative and potentially effective treatment of single or bilocular HCC and has been used for advanced-stage HCC as an alternative to TACE prior to be proposed as an alternate bridging therapy. SBRT is a high-precision technique allowing to deliver a precise treatment on moving lesions (integrating MRI technology) in a short time. While the radiosensitivity of the liver did not allow the use of conventional radiotherapy for patients on the waiting list for LT until several years ago, these new technical developments made it possible to administer hypofractionated external radiation more precisely. Therefore, this treatment modality is reported in patients with more advanced liver disease that would otherwise not have access to bridging therapy.

Advantages of SBRT, as compared to TACE or RF, are

* to preserve the hepatic artery, which can be altered by TACE
* to allow access to complex tumors locations or superficial lesions not feasible by RF
* to avoid any tumor spread related to punctures
* to avoid general anesthesia.

However, SBRT has not been validated as bridging therapy before LT in a prospective study. To date, data in the literature are heterogeneous, mostly based on retrospective studies and small patient number, and are not yet robust enough to pave the basement for a randomized trial comparing SBRT to the other bridging therapies for patients with HCC enlisted for LT. There is a lack of subgroup analyses of the role of SBRT in previously treated patients by ablation/surgery/TACE or naive patients (i.e.those in whom other bridge therapies are contraindicated) that could allow better clarification of SBRT indications as bridge therapy. It is also necessary to provide better understanding of imaging response after SBRT and its correlation with liver explant pathological response.

Succinct description of the intervention

SBRT is a high-precision technique allowing to deliver a precise high dose irradiation on moving lesions (integrating MRI technology) in a short time. While the radiosensitivity of the liver did not allow the use of radiotherapy for patients on the waiting list for LT until several years ago, these new technical developments made it possible to administer the external radiation more precisely. Patients will have 3 to 8 sessions delivered in one to three weeks. The overall duration is 3 weeks maximum.

Summary of the known and foreseeable benefits and risks for the research participants

Foreseable benefits are to provide access to a bridging therapy during waiting time for LT to patients who would not benefit otherwise from a bridging therapy. The objective is to prevent HCC progression during waiting time, which may result in drop-out from the waiting list and loss of access to a curative treatment.

Foreseable risks related to SBRT are toxicity which may be encountered during radiotherapy and which may be related to irradiation. Toxicity includes acute and late adverse side effects (from 6 months after the end of SBRT).).

Design of the study Prospective, single arm, multicentric, phase II trial according to a single stage A'Hern's design.

Number of participating sites Fifteen French LT centers trained in the technique of SBRT for HCC. Each LT center is paired with a radiation center.

Implementation of the study

Screening visit The screening visit will correspond to the multidisciplinary meeting evaluating LT indications and bridging therapy while waiting for LT for HCC patients in each LT center according to standard of care.

Inclusion visit and Baseline visit (D-30 to D-1 of the first SBRT session)

Information and informed consent Information about the study, along with usual information on LT, will be provided during a consultation by the surgeon or hepatologist then by the radiation oncologist to determine the final eligibility according to technical feasibility, and to explain the modalities, objectives and possible adverse effects of SBRT.

Final consent will be retrieved by the latest specialist seen by the patients before starting SBRT (usually the radiation oncologist).

Baseline visit (D-30 to D-1):

During this visit, a special attention will be paid to:

* Clinical examination: General performance status (PS) score, jaundice, ascites, encephalopathy.
* Calculation of Child-Pugh Score and MELD Score.
* Laboratory tests required (as done in usual care): baseline serum liver tests (ASAT, ALAT, gGT, PAL, albumin, bilirubin, PT, INR), serum alpha-foetoprotein, baseline blood count and platelets, baseline kidney function serum tests (creatinine, urea, Na, K).
* Paraclinical examinations required (usual care for HCC exploration): MRI liver imaging or Liver CT scan.

SBRT (M0)

Patients will have 3 to 8 sessions delivered in one to three weeks. The overall duration is 3 weeks maximum.

Patient' monitoring between the sessions will be in line with common practice.

Follow-up visits after the first session of SBRT and before LT (M1, M3, M6, M9, M12, M15 at maximum),

Liver transplantation (M15 at maximum)

Liver transplantation will be performed according to each center's usual practice. As the organ allocation is regulated on a national scale by the National Biomedecine Agency (ABM), patient's access to LT will be unchanged.

Data collected on standard operative report: intervention duration, blood loss amount, blood products transfusion, per-operative incidents, reconstruction modalities (arterial, portal, caval, biliary), reperfusion syndrome at declamping.

Data collected during post-LT hospital stay: occurrence of early complications (arterial, biliary, parietal, digestive, and other).

Data related to complications that may be related to SBRT will be recorded: biliary complications (fistulae/stenosis), arterial complications (stenosis), caval complications (haemorrhage/stenosis), delayed wound healing.

Post liver transplant follow up (maximum 39 months after inclusion and within 24 months post LT)

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* Patients enlisted for LT in France for HCC (under Agence de Biomédecine (ABM) regulation)
* HCC previously treated by ablation/surgery/TACE or naive
* Not suitable for another bridging therapy such as liver resection, ablation therapy, or TACE (discussed in multidisciplinary meeting within a transplant center)
* Suitable for stereotactic radiotherapy:
* ECOG, performance status score ≤ 2,
* Child-Pugh Score ≤ B7,
* Number of lesions between 1 and 3
* Maximum tumor size < 5cm Liver remnant volume ≥ 700 ml.
* Health insurance coverage.
* Written informed consent

Exclusion Criteria:

* Inability to comply with study procedures
* Patients under guardianship or curatorship
* Pregnancy (negative urinary/blood βHCG test)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 139 (Estimated)
Dates: Start 2024-05-31 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
To evaluate the efficacy of stereotactic body radiotherapy (SBRT) as bridging therapy for patients with hepatocellular carcinoma (HCC) enlisted for liver transplantation (LT). | Within 15 months following SBRT.
  Bridge therapy success is defined as follows:
  * Patient with liver transplantation within 15 months after the first session SBRT or,
  * Patient still enlisted (ie with aFP score<2) at M15 from the first session SBRT.
  All other cases will be considered as failure.

SECONDARY OUTCOMES:
To estimate the overall and disease-free survival after LT for HCC treated with SBRT on waiting list | Up to 24 months post LT
  * Overall survival (OS) at 39 months from SBRT among all patients treated with SBRT. OS is defined as the time from the first session of SBRT to death or last follow-up.
  * Disease free survival at 39 months from SBRT will be assessed among patients treated with SBRT and achieving the primary endpoint. DFS is defined as the time from the the first session of SBRT to CHC relapse or last follow-up.
To evaluate the pathological response after SBRT on the liver explant after LT | After LT surgery (maximum 39 months after inclusion and within 24 months post LT).
  Pathological response (necrosis rate and viable tumoral cells rate) on liver explant after LT
To assess the performance of liver imaging (using RECIST 1.1, mRECIST) to predict the pathological response | Preceding LT surgery (and within 15 months after inclusion at maximum)
  * Imaging response according to RECIST criteria (mRECIST and RECIST 1.1) assessed one month after the first session of SBRT and then every three months thereafter until LT
  * Correlation between the last imaging response before LT (mRECIST and RECIST 1.1) and the pathological response at LT.
To assess the occurrence of adverse events related to SBRT during waiting time period and after LT | Before and after LT (maximum 39 months after inclusion and within 24 months post LT)
  Adverse events possibly related to SBRT:
  * on waiting list: radiation induced liver disease (Calculation of MELD-score and Child-Pugh score every 3 months), radiation pneumonitis (imaging evaluation every 3 months)
  * per-operative events during LT (in particular, technical issues for vascular and biliary reconstructions due to tissue frailty)
  * post-operative complications rate (vascular and biliary complications, post-LT liver failure, pulmonary decompensation).

CONTACTS AND LOCATIONS:
Overall Officials: Claire GOUMARD, MD, PhD Assistant Professor, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Service de chirurgie digestive, hépato-bilio-pancréatique et transplantation hépatique. Groupe Hospitalier Pitié-Salpêtrière, Paris, France

IPD SHARING:
Plan to Share IPD: No